CLINICAL TRIAL: NCT04465266
Title: A Phase 1 Crossover Study of Single and Multiple Dose Pharmacokinetics, and Dose Linearity, of Tolperisone in Healthy Subjects
Brief Title: A Phase 1 PK Study of Tolperisone in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurana Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CLN-110
Record Dates: First submitted 2020-07-02; First posted 2020-07-10 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Healthy
MeSH Terms: interventions — Tolperisone

STUDY DESIGN:
Intervention Model Description: sequence randomized
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 50 mg Tolperisone (Experimental): 50 mg tablets (2 days SD, 2 days TID)
  Interventions: Drug: Tolperisone
- 100 mg of Tolperisone (Experimental): 100 mg tablets (2 days SD, 2 days TID)
  Interventions: Drug: Tolperisone
- 200 mg Tolperisone (Experimental): 200 mg tablets (2 days SD, 2 days TID)
  Interventions: Drug: Tolperisone

INTERVENTIONS:
Drug: Tolperisone — tablets

SUMMARY:
This is a randomized, single-blind, single and multiple dose crossover subjects in healthy adult subjects

DETAILED DESCRIPTION:
This is a single-center, in-patient, treatment sequence-randomized, single-blind SD and MD crossover study in 27 healthy adult male and female subjects. Subjects will be admitted to the clinic on Day-1 and discharged the morning of Day 5 of each treatment period. Subjects will be on a standard diet during each inpatient treatment period; study drug will be administered in the fasted state for PK assessments on Days 1 and 4 of each treatment period. Subjects will have a follow-up phone call 7 to 10 days after the last dose in Period 3. There will be a 6 to 8 day washout between the last dose in Period 1 and the first dose in Period 2, and between the last dose in Period 2 and the first dose in Period 3.

ELIGIBILITY:
Inclusion Criteria:

* Generally Healthy Subjects
* BMI between 18.5 and 32.5 kg/m2

Exclusion Criteria:

- pregnant or breastfeeding

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Cmax | taken over 4 days per dose
  Maximum plasma concentration of tolperisone
Tmax | taken over 4 days per dose
  Time of maximum plasma concentration of tolperisone
AUC | taken over 4 days per dose
  Area under the curve of tolperisone plasma concentrations
T1/2 | taken over 4 days per dose
  Half life of tolperisone

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials Early Phase Services, LLC, San Antonio, Texas, United States